CLINICAL TRIAL: NCT07390890
Title: Efficacy of Direct Selective Laser Trabeculoplasty (DSLT) for Reducing Medication Burden in Medically Controlled Patients With Ocular Hypertension or Primary Open Angle Glaucoma
Brief Title: DSLT for Reducing Medication in Glaucoma
Status: Recruiting | Type: Observational
Sponsor: The Eye Institute of West Florida (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: ND-25-01
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Voyager DSLT — Voyager DSLT

SUMMARY:
This is a prospective, single arm, open label study conducted at a single site to evaluate the efficacy of Direct Selective Laser Trabeculoplasty (DSLT) in reducing medication burden in patients with medically controlled ocular hypertension or primary open angle glaucoma.

The study will assess the primary endpoint of reduction in medication count at 6 months compared to baseline. Secondary endpoints include IOP reduction compared to baseline (both percentage and absolute), complete success rate (no increase in IOP without medications), proportion of eyes needing medication at 6 months, and any secondary surgical interventions at 6 months post-DSLT.

Participants will undergo DSLT with 120 shots, 400 µm spot size, and 1.8mJ fixed energy delivered at the limbus over 2.4 seconds. Follow-up visits will occur at 1 month, 3 months, and 6 months post-procedure, with IOP measured using a calibrated Goldmann tonometer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled to undergo DSLT treatment in one or both eyes.

  * Diagnosis of ocular hypertension or primary open angle glaucoma (POAG).
* Medically controlled on 1-3 topical ocular hypotensive agents with IOP ≤21 mmHg.

Exclusion Criteria:

* Previous glaucoma surgeries/interventions:

  * Patients who have undergone prior glaucoma-related procedures (e.g., trabeculectomy, laser trabeculoplasty, MIGS, or tube shunt).
* Patients who have undergone cataract surgery within the prior 2 years.
* Secondary glaucoma:

  * Patients with secondary forms of glaucoma, such as angle-closure glaucoma, neovascular glaucoma, or glaucoma resulting from trauma or other systemic diseases.
* Other significant ocular conditions including advanced cataracts, retinal diseases (e.g., age-related macular degeneration), or any condition that might complicate the assessment of intraocular pressure (IOP) or visual function as deemed by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with ocular hypertension or POAG undergoing DSLT treatment in one or both eyes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2027-01-26 (Estimated); Study Completion 2027-01-26 (Estimated)

PRIMARY OUTCOMES:
Reduction in the number of glaucoma medications required to maintain target intraocular pressure (IOP) | 6 months post-DSLT treatment
  The primary outcome will be assessed by comparing the number of medications needed to maintain target IOP before and after DSLT treatment.

SECONDARY OUTCOMES:
Change in intraocular pressure (IOP) from baseline | 6 months post-DSLT treatment
  IOP will be measured using Goldmann applanation tonometry at each follow-up visit.
Proportion of eyes needing medication stratified by number of IOP medications required | 6 months post-DSLT treatment
Number and type of Secondary surgical interventions | 6 months post-DSLT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Neel Desai, MD, Principal Investigator — The Eye Institute of West Florida
Locations (1):
- The Eye Institute of West Florida, Largo, Florida, United States